CLINICAL TRIAL: NCT02442206
Title: A Randomized, Double-blinded, Single-center, Placebo Controlled, Cross-over Study to Assess the Effect of QVA149 (Indacaterol Maleate / Glycopyrronium Bromide) on Cardiac Function in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effect of QVA149 (Indacaterol Maleate/Glycopyrronium Bromide) on Cardiac Function in COPD Patients
Acronym: CLAIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149ADE05; 2014-004680-21 (EudraCT Number)
Record Dates: First submitted 2015-05-06; First posted 2015-05-13 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
Keywords: QVA149, cardiac function, ventricular enddiastolic volume, hyperinflated COPD patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1 (Experimental): QVA149 from day 1 to day 15 followed by Placebo from day 29 to day 43
  Interventions: Drug: QVA149; Drug: Placebo
- Treatment sequence 2 (Experimental): Placebo from day 1 to day 15 followed by QVA149 from day 29 to day 43
  Interventions: Drug: QVA149; Drug: Placebo

INTERVENTIONS:
Drug: QVA149 — QVA149 capsules 100/50 µg for inhalation via Concept-1-inhaler, taken once daily
  Other Names: Ultibro
Drug: Placebo — Placebo to QVA140 capsules 100/50 µg for inhalation via Concept-1-inhaler, taken once daily

SUMMARY:
This mechanistic study is a single-center, randomized, double-blind, placebo-controlled, cross-over study to evaluate the effect of dual bronchodilation with QVA149 on cardiac and lung function parameters in hyperinflated COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with airflow limitation indicated by a post-bronchodilator FEV1 <80% of the predicted normal value and a post-bronchodilator FEV1/FVC<0.7
* Current or ex-smokers who have a smoking history of at least 10 pack years.
* Able and willing to give written informed consent
* Hyperinflated patients with RVol>135% predicted

Exclusion Criteria:

* Patients on LABA or LAMA treatment at Visit 1.
* History of one COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization 3 months prior to Visit 2.
* More than one COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization within 6 months prior to Visit 2.
* Patients who have clinically significant cardiovascular abnormalities, which could interfere with the assessment of the study treatment (such as but not limited to cardiac arrhythmias, heart failure with left ventricular ejection fraction <40% as determined by MRI scan, unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, history of myocardial infarction 6 months prior to Visit 2)
* Patients with a known history or current atrial fibrillation to be confirmed by ECG.
* Patients with pacemaker, bypass or stent.
* Patients whose QTcF measured at Visit 3 is >450 ms for males and >470 ms for females

Additional study-specific inclusion and exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Hanover, Germany

REFERENCES:
- [Derived] Vogel-Claussen J, Schonfeld CO, Kaireit TF, Voskrebenzev A, Czerner CP, Renne J, Tillmann HC, Berschneider K, Hiltl S, Bauersachs J, Welte T, Hohlfeld JM. Effect of Indacaterol/Glycopyrronium on Pulmonary Perfusion and Ventilation in Hyperinflated Patients with Chronic Obstructive Pulmonary Disease (CLAIM). A Double-Blind, Randomized, Crossover Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1086-1096. doi: 10.1164/rccm.201805-0995OC. PMID 30641027
- [Derived] Hohlfeld JM, Vogel-Claussen J, Biller H, Berliner D, Berschneider K, Tillmann HC, Hiltl S, Bauersachs J, Welte T. Effect of lung deflation with indacaterol plus glycopyrronium on ventricular filling in patients with hyperinflation and COPD (CLAIM): a double-blind, randomised, crossover, placebo-controlled, single-centre trial. Lancet Respir Med. 2018 May;6(5):368-378. doi: 10.1016/S2213-2600(18)30054-7. Epub 2018 Feb 21. PMID 29477448

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 30 | 32
Completed | 29 | 29
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 1
Not completed — withdrew consent | 0 | 1
Not completed — COPD exacerbation | 0 | 1
Period: Period 2
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 29 | 29
Completed | 28 | 29
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.00) | 63.8 (7.80) | 63.9 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 22 | 23 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 32 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End-diastolic Volume (LVEDV)
Description: Left ventricular enddiastolic volume (LVEDV) is a measurement of the volume of blood in the heart's left ventricular chamber at the end of the chamber's filling with blood and will be determined as measured by MRI.
Time Frame: Baseline, week 2
Population: Per protocol set (PPS) included all patients in the FAS who did not have any major protocol deviations. Only patients with a valid LV EDV value at both baseline and post-baseline in a period were included
Measure: Mean (Standard Deviation); unit: ML
Groups:
- QVA149: QVA149 from day 1 to day 15 followed by Placebo from day 29 to day 43
- Placebo: Placebo from day 1 to day 15 followed by QVA149 from day 29 to day 43
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
ML | 11.873 (14.3215) | -0.954 (12.2463)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = 10.270, 95% CI 2-sided [6.209 to 14.331]

2. Secondary Outcome: Change in Forced Expiratory Volume in One Second (FEV1).
Description: Forced Expiratory Volume in one second (FEV1) will be calculated as the volume of air forcibly exhaled in one second as measured by spirometry.
Time Frame: Baseline, week 2
Population: Per protocol set (PPS) included all patients in the FAS who did not have any major protocol deviations. Only patients with a valid value for parameter at both baseline and post-baseline in a period are included - Period baseline was defined as the value taken in each period prior to start of study treatment
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Liter | 0.42 (0.211) | -0.01 (0.168)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = 0.42, 95% CI 2-sided [0.36 to 0.49]

3. Secondary Outcome: Change in Forced Vital Capacity (FVC).
Description: Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC will be assessed via spirometry.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Liter | 0.67 (0.434) | 0.00 (0.293)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = 0.67, 95% CI 2-sided [0.55 to 0.80]

4. Secondary Outcome: Change in Inspiratory Capacity (IC) at Each Time-point
Description: Inspiratory capacity (IC) was defined as the mean of the maximum IC over 3 values measured by bodyplethysmography according to internationally accepted standards.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Liters | 0.475 (0.3284) | 0.014 (0.2388)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = 0.446, 95% CI 2-sided [0.352 to 0.541]

5. Secondary Outcome: Change in Total Lung Capacity (TLC)
Description: Total Lung Capacity (TLC) will be calculated from the mean Functional Residual Capacity (FRC) plus the highest value of the Inspiratory Capacity, both measured by body plethymography according to internationally accepted standards.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Liters | -0.181 (0.3408) | -0.001 (0.3618)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p = 0.0017, ANOVA; Mean Difference (Net) = -0.177, 95% CI 2-sided [-0.285 to -0.070]

6. Secondary Outcome: Change in Residual Volume (RVol)
Description: Residual Volume (RVol) will be calculated from the value of Total Lung Capacity (TLC) minus the highest value of the Slow Vital Capacity, both measured by body plethymography according to internationally accepted standards.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Liters | -0.757 (0.5833) | 0.012 (0.5141)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -0.751, 95% CI 2-sided [-0.925 to -0.577]

7. Secondary Outcome: Change in Specific Airway Resistance (sRaw)
Description: Specific Airway Resistance (sRaw) will be documented as effective resistance (sReff) calculated as the median of five acceptable measurements. Values will be measured by body plethymography according to internationally accepted standards.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kPa*s/L
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 56 | 55
kPa*s/L | -1.887 (1.0979) | 0.037 (1.0383)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -1.639, 95% CI 2-sided [-1.945 to -1.332]

8. Secondary Outcome: Change in Functional Residual Capacity (FRC)
Description: Functional Residual Capacity (FRC) will be calculated as the mean of three reproducible values as measured by body plethymography according to internationally accepted standards.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Liters | -0.656 (0.4602) | -0.015 (0.4257)
Statistical Analysis 1: Comparison: QVA149; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Net) = -0.625, 95% CI 2-sided [-0.761 to -0.489]

9. Secondary Outcome: Change in Right Ventricular (RV) and Left Ventricular (LV) Ejection Fraction (EF)
Description: Right and left ventricular ejection fraction is the fraction of blood (in percent) pumped out of the heart's left and right ventricular chamber, respectively, with each heart beat and will be determined as measured by MRI.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Percentage
  LV-EF: number analyzed (Participants) | 56 | 54
  LV-EF | 1.893 (5.8486) | 1.313 (5.4261)
  RV-EF: number analyzed (Participants) | 56 | 54
  RV-EF | 2.046 (5.8746) | 0.361 (6.1936)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; LV EF; Test type: Superiority; p = 0.1420, ANOVA; Mean Difference (Net) = 1.209, 95% CI 2-sided [-0.419 to 2.836]
Statistical Analysis 2: Comparison: QVA149 vs Placebo; RV EF; Test type: Superiority; p = 0.1732, ANOVA; Mean Difference (Net) = 1.131, 95% CI 2-sided [-0.512 to 2.774]

10. Secondary Outcome: Change in Left and Right Ventricular End-systolic Volume
Description: Right ventricular end-systolic volume (RV-ESV) and left ventricular end-systolic volume (LV-ESV) is a measurement of the volume of blood in the heart's right and left ventricular chamber, respectively, at the end of the heart's contraction and will be determined as measured by MRI.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ML
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
ML
  LV-ESV: number analyzed (Participants) | 56 | 54
  LV-ESV | 1.898 (8.4565) | -2.283 (8.1489)
  RV-ESV: number analyzed (Participants) | 56 | 54
  RV-ESV | 2.183 (8.7063) | 0.133 (9.3370)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; LV ESV; Test type: Superiority; p = 0.0437, ANOVA; Mean Difference (Net) = 2.241, 95% CI 2-sided [0.066 to 4.417]
Statistical Analysis 2: Comparison: QVA149 vs Placebo; RV ESV; Test type: Superiority; p = 0.1236, ANOVA; Mean Difference (Net) = 2.095, 95% CI 2-sided [-0.591 to 4.782]

11. Secondary Outcome: Change in Right Ventricular Enddiastolic Volume
Description: Right ventricular end-diastolic volume is a measurement of the volume of blood in the heart's right ventricular chamber at the end of the chamber's filling with blood and will be determined as measured by MRI.
Time Frame: Baseline, week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ML
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
ML | 12.323 (13.9683) | 1.758 (14.7904)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; Test type: Superiority; p = 0.0002, ANOVA; Mean Difference (Net) = 9.357, 95% CI 2-sided [4.649 to 14.065]

12. Secondary Outcome: Cardiac Output at Each Time-point, Left and Right Ventricular Cardiac Output (LVCO and RVCO)
Description: Cardiac output is calculated as the heart rate multiplied by the stroke volume (= difference between ventricular enddiastolic volume and endsystolic volume) that will be determined as measured by MRI.
Time Frame: week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liter/min
Arm/Group | QVA149 | Placebo
Number analyzed (Participants) | 57 | 59
Liter/min
  LVCO: number analyzed (Participants) | 56 | 54
  LVCO | 0.504 (0.7919) | 0.119 (0.8970)
  RVCO: number analyzed (Participants) | 56 | 54
  RVCO | 0.517 (0.8063) | 0.144 (0.9523)
Statistical Analysis 1: Comparison: QVA149 vs Placebo; LVCO; Test type: Superiority; p = 0.0032, ANOVA; Mean Difference (Net) = 0.337, 95% CI 2-sided [0.118 to 0.555]
Statistical Analysis 2: Comparison: QVA149 vs Placebo; RVCO; Test type: Superiority; p = 0.0182, ANOVA; Mean Difference (Net) = 0.281, 95% CI 2-sided [0.050 to 0.512]

ADVERSE EVENTS:
Time Frame: For the study duration of about 13 weeks
Groups:
- QVA149 (110/50): QVA149 (110/50)
- Placebo: Placebo
- All Patients: All Patients
Arm/Group | QVA149 (110/50) | Placebo | All Patients
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/61 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/59 | 2/61 | 2/62
Other Adverse Events (participants affected / at risk) | 27/59 | 17/61 | 40/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (110/50) (N=59) | Placebo (N=61) | All Patients (N=62)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (110/50) (N=59) | Placebo (N=61) | All Patients (N=62)
Vertigo (Ear and labyrinth disorders) | 3 | 3 | 6
Nasopharyngitis (Infections and infestations) | 3 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Headache (Nervous system disorders) | 4 | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-11-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02442206/SAP_000.pdf
  • Study Protocol (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02442206/Prot_001.pdf